CLINICAL TRIAL: NCT01452035
Title: Comparing the Effects Exercise Intensity and Energy Expended During a Single Exercise Session on Insulin Sensitivity and Fatty Acid Partitioning Within Skeletal Muscle the Next Day in Obese Adults.
Brief Title: Exercise Dose Response for Improving Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Associate Professor, Movement Science, School of Kinesiology, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R01 DK077966 - MX; R01DK077966 (NIH)
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Obesity
Keywords: insulin sensitivity; fatty acid metabolism; exercise
MeSH Terms: conditions — Obesity; Insulin Resistance; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental)
  Interventions: Other: Exercise
- Sedentary Control (No Intervention)

INTERVENTIONS:
Other: Exercise — single session of exercise
  Arms: Exercise

SUMMARY:
Many of the beneficial metabolic effects of endurance exercise training are not due to adaptations to weeks, months, or even years of training, but rather much is due to the response to the most recent exercise session(s). Therefore, the investigators contend that lifestyle interventions for obese individuals should be tailored to optimize the metabolic effects of the most recent exercise session(s). But the "dose" of exercise necessary to evoke these beneficial responses is not known, and the mechanisms responsible for these improvements are poorly understood. The findings from these studies will: 1) establish the minimum "dose" of a single exercise session necessary to improve insulin sensitivity the next day in obese adults, 2) characterize the underlying metabolic factors responsible for the improvement in insulin sensitivity, and 3) assess the cumulative metabolic adaptations that occur over days, weeks, and months of a low-intensity/low-volume lifestyle exercise program. Findings from these studies will provide valuable information for the development of lifestyle programs aimed at maximizing the key metabolic health benefits of each exercise session in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index [BMI] = 30-45 kg/m2, weight stable (± 5 lbs in the past month), fasting blood glucose concentration must be <125 mg/dl.

Exclusion Criteria:

* pregnancy, evidence of cardiovascular or metabolic disease, taking medications know to influence metabolism.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2009-01; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | 2-3 hours
  A hyperinsulinemic-euglycemic clamp will be used to assess peripheral insulin sensitivity and will be performed using a primed 2h insulin infusion at a rate of 100 mU/m2/min.

SECONDARY OUTCOMES:
Resting Metabolic Rate | 40-60 min
Meal Tolerance Test | 2-3h

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Horowitz, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- Michigan Clincal Research Unit, Ann Arbor, Michigan, United States